CLINICAL TRIAL: NCT03054480
Title: A Comparative Study for Efficacy and Safety Between Fractional Micro-Needle Radiofrequency (FRM) and Intradermal Botulinum Toxin A for the Treatment of Primary Axillary Hyperhidrosis
Brief Title: Fractional Micro-Needle Radiofrequency and I Botulinum Toxin A for Primary Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Thep Chalermchai, Principal Investigator, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 109/1-59
Record Dates: First submitted 2017-02-11; First posted 2017-02-15 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Primary Axillary Hyperhidrosis
Keywords: Fractional Micro-Needle Radiofrequency; Intradermal Botulinum Toxin A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional Micro-Needle Radiofrequency (Experimental): each patient will be treated with FMR DeAge®, applicator device at 4-week intervals for 2 sessions of treatment. This applicator consists of rows of 36 (6x6 needles) insulated microneedles that form an array of positively and negatively charged electrodes. The microneedles will deliver bipolar radiofrequency energy in a fractional manner that extends from 3.0 mm below the surface of the skin. All subjects will be prepared by local anesthesia to induce numbness at the axilla prior to treatment. The targeted axillary side will be treated with a total of 4 passes.
  Interventions: Device: Fractional Micro-Needle Radiofrequency
- Botulinum toxin type A (Active Comparator): 50 units of Botulinum toxin type A will be intradermal injected over axillary area. The protocol by using 1-2 units per 1 injection area with the coverage of 1x1 cm2 will be treated.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Device: Fractional Micro-Needle Radiofrequency
  Other Names: DeAgeEX Fractional RF
  Arms: Fractional Micro-Needle Radiofrequency
Drug: Botulinum toxin type A
  Other Names: Neuronox
  Arms: Botulinum toxin type A

SUMMARY:
Because of the limiting data about an efficacy and safety of fractional radiofrequency for the treatment of hyperhidrosis, this study aim to compare clinical efficacy by Hyperhidrosis Disease Severity Score (HDSS) between Fractional Microneedle Radiofrequency device and intradermal Botulinum toxin type A injection for the treatment of primary axillary hyperhidrosis. The secondary objectives to determine the improvement change of iodine starch test, total amount of sweat production by trans-epidermal water loss (TEWL), patient's satisfaction and their quality of life by Dermatology Life Quality Index and side effect between the groups.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects, age between 18-60 years

* Healthy volunteers
* Subjects who have experienced with excessive sweating on both sides of axillary areas and have a positive result for iodine starch test on the screening day
* Willing to participant into the study and voluntary to sign in the informed consent form

Exclusion Criteria:

Active bacterial or fungal infection over tested area / axillae

* Pregnancy and breast feeding
* Previously underwent the surgical treatment such as radical resection of sweat glands for primary axillary hyperhidrosis
* Currently being treated with intradermal botulinum toxin type A injection at axillary area for less than 12 months
* Currently being inserted the cardiac pace maker or any other internal electronic devices
* Secondary hyperhidrosis caused by hyperthyroidism, drug induced, abnormal autonomic or neurological disorder that affect sweat gland
* Allergy to botulinum toxin type A
* Known contact allergy to iodine
* Unable to follow and comply to the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
The change of Hyperhidrosis disease severity score (HDSS) at week-12 with the baseline | 12 weeks
  Hyperhidrosis disease severity score will be assessed by study subjects that is categorized to 4 levels; (1) my axillary sweating is never noticeable and never interferes with my daily activities (2) my axillary sweating is tolerable but sometimes interferes with my daily activities (3) my axillary sweating is barely tolerable and frequently interferes with my daily activities (4) my axillary sweating is intolerable and always interferes with my daily activities

SECONDARY OUTCOMES:
Iodine starch test | baseline, week 4 and week 12
  Qualitative test used to evaluate sudo-motor function (sweating) which method is to apply iodine solution to the skin. Once dry, the area is dusted with cornstarch or potato flour then sweating is encouraged. When sweat reaches the surface of the skin the starch and iodine combine causing a dramatic color change from yellow to dark blue allowing sweat production to be actively visualized.
  Photograph from iodine starch test will be assessed by two independent clinical assessors who are blinded to study protocol and grading with score. The investigators will prepare the photo with pre- and post-treatment set. Each set will contain 6 photos, 3 photos from the left and 3 photos from the right. Prepare by using Microsoft PowerPoint program, on each slide will contain 2 photos, pre-treatment photos on the left and post treatment photos on the right. The paired photos will be assessed and graded the score at different time points (4 and 12 weeks) on each side of axilla
Participants' satisfaction assessment | week 4 and week 12
  An assessment will be determined at the endpoint visit (4th-12thweek) after the treatment by study subjects by Quartile rating scale on each side of axilla. Quartile rating scale by comparing with the baseline that is categorized to 4 levels; (3) greatly satisfy with treatment result (2) moderately satisfy with treatment result (1) slightly satisfy with treatment result (0) No different with treatment result.
Adverse effect | 12 weeks
  Side effect

IPD SHARING:
Plan to Share IPD: No